CLINICAL TRIAL: NCT05407974
Title: Pleurectomy Versus Pleural Abrasion in Patients With Spontaneous Pneumothorax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pleurectomy Versus abrasion
Record Dates: First submitted 2022-04-05; First posted 2022-06-07 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleural abrasion Group (Experimental): Mechanical pleural abrasion will be performed by rubbing the parietal pleura with gauze or a cleaning pad.
  Interventions: Procedure: pleurectomy
- pleurectomy group (Experimental): Pleurectomy will be performed by a small piece of gauze on grasper. The aim of pleurectomy is to remove the parietal pleural especially above the areas with blebs or bullae.
  Interventions: Procedure: pleurectomy

INTERVENTIONS:
Procedure: pleurectomy — All patients will undergo resection of apical blebs with simultaneous pleurectomy or pleural abrasion.
  Chest tube will be inserted in the pleural cavity and maybe connected on low-grade suction for first 24 h according to type of pneumothorax & surgeons' preference, after which the suction is disconnected.
  Post Operatively both groups will be compared regarding the postoperative drainage amount, persistence of air leak (chest tube removal time), length of hospital stay, mortality and risk of recurrence.
  Follow up Chest x-ray will be done immediate postoperatively, then each patient will be followed up after 6 months.
  Other Names: bullectomy

SUMMARY:
Pneumothorax refers to air in the pleural cavity (i.e. interspersed between the lung and the chest wall).1 Primary spontaneous pneumothorax (PSP) mostly occurs in healthy individuals without an apparent cause, probably due to the rupture of subpleural blebs located mostly on the apex of the lung or the apical segment of the lower lobe. Compared to PSP, a secondary spontaneous pneumothorax (SSP) occurs in the setting of underlying pulmonary disease, like COPD.2 Surgical treatment involves resection of apical bleb disease and pleurodesis which could be chemical or mechanical. Mechanical pleurodesis accomplished either via pleurectomy or pleural abrasion.3 In this study, we aim to compare the efficiency and recurrence risk of pleural abrasion versus pleurectomy in patients with Spontaneous pneumothorax.

DETAILED DESCRIPTION:
Pneumothorax is a relatively common clinical problem which can occur in individuals of any age. Irrespective of aetiology (primary, or secondary to lung disorders or injury), immediate management depends on the extent of cardiorespiratory impairment, degree of symptoms and size of pneumothorax. 4 The presentation of a pneumothorax varies between minimal pleuritic chest discomfort and breathlessness to a life threatening medical emergency with cardiorespiratory collapse requiring immediate intervention.5-7 Typical signs include reduced breath sounds, reduced ipsilateral chest expansion and hyper resonant percussion note. Mediastinal shift away from the affected side, tachycardia, tachypnea and hypotension occur in Tension pneumothorax. 8 Pneumothorax can be categorized as spontaneous which maybe primary or secondary and traumatic according to aetiology. Occasionally, individuals may develop a concomitant haemothorax due to bleeding caused by shearing of adjacent subpleural vessels when the lung collapses.4 A primary spontaneous pneumothorax (PSP) is a condition that occurs predominantly in young and thin male individuals who do not have any history of underlying lung disease. Although it is mostly attributed to the rupture of a subpleural bleb or bulla, the exact cause of PSP is still unknown.1 Moreover, current cigarette smoking greatly increases the risk of developing PSP by as much as nine times, with evidence of a dose-response relationship.9 Secondary spontaneous pneumothorax (SSP) frequently occurs in association with primary diseases, such as chronic obstructive pulmonary disease (COPD), interstitial pneumonia (IP), and pulmonary fibrosis disease (PFD). 10 Treatment of spontaneous pneumothorax depends on the patient's condition and can range from conservative treatment, drainage, and pleurodesis, to surgical treatment.10 Surgical treatment is based on resection of bullous lesions causing air leakage and techniques to prevent recurrence. Surgical treatment without additional pleurodesis may increase the risk of recurrence, Various pleurodesis techniques such as chemical pleurodesis or mechanical pleurodesis via pleural abrasion or pleurectomy are used to reduce the recurrence rate.1

ELIGIBILITY:
Inclusion Criteria:

* - Patients presented with spontaneous pneumothorax; primary or secondary.
* Age: all age groups are included
* Approach: Video assisted thoracoscopic surgery

Exclusion Criteria:

* - Refusal of procedure or participation in the study.
* Patients with acquired pneumothorax (eg. Traumatic)
* Patients with history of previous thoracic surgery on the same side of chest.
* Approach: any open thoracotomy approach or switching from VATS to open thoracotomy

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-03 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Recurrence | 6 months
  Incidence of recurrence of pneumothorax is measured by clinical examination and chest x ray done at 3 and at 6 month postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Abdelfatah E Abugabal, Principal Investigator — Ainshams University
Locations (1):
- Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ocakcioglu I, Kupeli M. Surgical Treatment of Spontaneous Pneumothorax: Pleural Abrasion or Pleurectomy? Surg Laparosc Endosc Percutan Tech. 2019 Feb;29(1):58-63. doi: 10.1097/SLE.0000000000000595. PMID 30499890
- [Background] Henry M, Arnold T, Harvey J; Pleural Diseases Group, Standards of Care Committee, British Thoracic Society. BTS guidelines for the management of spontaneous pneumothorax. Thorax. 2003 May;58 Suppl 2(Suppl 2):ii39-52. doi: 10.1136/thorax.58.suppl_2.ii39. No abstract available. PMID 12728149
- [Background] Joharifard S, Coakley BA, Butterworth SA. Pleurectomy versus pleural abrasion for primary spontaneous pneumothorax in children. J Pediatr Surg. 2017 May;52(5):680-683. doi: 10.1016/j.jpedsurg.2017.01.012. Epub 2017 Jan 27. PMID 28168984